CLINICAL TRIAL: NCT02107378
Title: A Randomized, Open-label, Parallel Group, Multi-center Phase II Clinical Trial Evaluating Effect of Addition of DCVAC/OvCa to Standard Chemotherapy in Women With Relapsed Platinum (Pt)-Resistant Epithelial Ovarian Carcinoma
Brief Title: Efficacy of DCVAC/OvCa Plus Standard of Care in Relapsed Platinum Resistant Epithelial Ovarian Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOV03
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-01

CONDITIONS: Epithelial Ovarian Carcinoma
Keywords: Immunotherapy; Serous; Relapsed; Platinum resistant (pt); Ovarian Cancer (OvCa); Biological; Vaccine
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Recurrence; Ovarian Neoplasms | interventions — Standard of Care; Paclitaxel; Topotecan; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCVAC/OvCa in parallel with chemo (SoC) (Experimental): Combination therapy with DCVAC/OvCa and Standard of Care (SoC)
  Interventions: Biological: DCVAC/OvCa
- Standard of Care (Chemotherapy) (Active Comparator): Standard of Care as an Active Comparator (Paclitaxel or topotecan or doxorubicin is Standard of Care First Line Chemotherapy)
  Interventions: Drug: Standard of Care (Paclitaxel or topotecan or doxorubicin)

INTERVENTIONS:
Biological: DCVAC/OvCa — DCVAC/OvCa is the experimental therapy added on to Paclitaxel or topotecan or doxorubicin
  Arms: DCVAC/OvCa in parallel with chemo (SoC)
Drug: Standard of Care (Paclitaxel or topotecan or doxorubicin) — Paclitaxel or topotecan or doxorubicin is Standard of Care First Line Chemotherapy
  Other Names: Paclitaxel; topotecan; doxorubicin
  Arms: Standard of Care (Chemotherapy)

SUMMARY:
The purpose of this study is to determine whether DCVAC/OvCa added to chemotherapy may result in prolongation of Overall Survival (OS).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether DCVAC/OvCa added to Standard of Care chemotherapy may result in prolongation of Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years or older
* Histologically confirmed International Federation of Gynecology and Obstetrics (FIGO) Stage III or IV epithelial ovarian, primary peritoneal, or fallopian tube carcinoma (serous, endometrioid or mucinous), who have undergone initial surgery or interval debulking surgery but have not reached complete remission of more than 6 months after first line platinum based chemotherapy, for one of the following reasons
* Patients are platinum-refractory (no response)
* Complete remission was not reached (partial responders)
* Relapse within ≤6 months of remission (Platinum-resistant)
* Platinum-based chemotherapy failure should have been confirmed by computerized tomography (CT)/magnetic resonance imaging (MRI) scan (Platinum-resistant) or by finding described as 'did not reach complete clinical remission' (Platinum-refractory or Platinum-partial response) Patients must have at least one measureable target lesion as defined by the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2

Exclusion Criteria:

* FIGO I,II epithelial ovarian cancer
* FIGO III, IV clear cells epithelial ovarian cancer
* Non-epithelial ovarian cancer
* Borderline tumors (tumors of low malignant potential)
* Prior or current systemic anti-cancer therapy for ovarian cancer [for example chemotherapy, monoclonal antibody therapy, tyrosine kinase inhibitor therapy, vascular endothelial growth factor (VEGF) therapy or hormonal therapy] except first line Platinum-based chemotherapy (with or without bevacizumab)
* Previous radiotherapy to the abdomen and pelvis
* Malignancy other than epithelial ovarian cancer, except those that have been in clinical remission (CR) for a minimum of 3 years, and except carcinoma in-situ of the cervix or non-melanoma skin carcinomas
* Clinically significant cardiovascular disease
* Active autoimmune disease requiring treatment
* History of severe forms of primary immune deficiencies
* Systemic immunosuppressive therapy for any reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Overall survival (all cause mortality) | 72 weeks

SECONDARY OUTCOMES:
Progression Free Survival | 72 weeks
  Per modified RECIST
Objective Response Rate | 0, 8, 16, ,24, 32, 40, 48, 56, 64, 72 weeks
  Per RECIST
Biological Progression Free Interval | 0, 8, 16, 24, 32, 40, 48, 56, 64, 72 weeks
Immunological Response | 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 weeks
Frequency of Adverse Events | 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 48, 56, 64, 72 weeks
Evaluation of Quality of Life via Functional Assessment of Cancer Therapy-Ovarian | 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 48, 56, 64, 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ales Horacek, Study Director — Accord Research
Locations (12):
- Czechia (5):
  - Brno
  - Nový Jičín
  - Olomouc
  - Ostrava
  - Prague
- Germany (3):
  - Cologne
  - Dresden
  - Erlangen
- Poland (4):
  - Bialystok
  - Krakow
  - Lublin
  - Poznan

IPD SHARING:
Plan to Share IPD: Undecided